CLINICAL TRIAL: NCT05160298
Title: Analgesic Effect of Bilateral Erector Spinae Plane Block With Ropivacaine After Sternotomy in Cardiac Surgery
Brief Title: Analgesic Effect of Bilateral Erector Spinae Plane Block With Ropivacaine After Sternotomy for Cardiac Surgery
Acronym: ESB-Sterno
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESB-Sterno (RBHP2021ELJEZI)
Record Dates: First submitted 2021-10-18; First posted 2021-12-16 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Cadiac Surgery; Median Sternotomy; Regional Anesthesia; Postoperative Pain
Keywords: Postoperative analgesia; Erector spinae plane block; Local anesthetics; Ropivacaine; Sternotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: * The ropivacaine group (42 patients): Echo-guided bilateral erector spinae block at the arrival in the intensive care unit. 20ml of Ropivacaine 2mg/ml for each side.
  * The control group (42 patients): Sham block bilaterally.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient will be under sedation during the block performance. Th nurse in charge to the patient will be absent during the block performance and the block will be realized by the practitioner who will not take care of the patient during his hospitalization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine group (Experimental): Performance of an echo-guided bilateral erector spinae block at the arrival in the intensive care unit with 20ml of Ropivacaine 2mg/ml in each side.
  Interventions: Drug: Ropivacaine 0,2% Injectable Solution
- Control group (Sham Comparator): Performance of a sham block at the arrival in the intensive care unit with no drugs administration
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Ropivacaine 0,2% Injectable Solution — Echo-guided bilateral erector spinae block
  Arms: Ropivacaine group
Other: Control group — Sham block
  Arms: Control group

SUMMARY:
The sternotomy site is the most painful area after cardiac surgery. Erector spinae plane block is effective in thoracic and abdominal surgery, but literature is lacking in cardiac surgery. The bilateral erector spinae plane block could reduce pain at rest and during mobilization, reduce opioids consumption, decrease postoperative complications, improve respiratory outcomes and improve patient comfort and satisfaction. The research hypothesis is that a single shot bilateral erector spinae plane block could reduce pain during mobilization during the first 48 hours after cardiac surgery performed with sternotomy

DETAILED DESCRIPTION:
Background:

Pain after cardiac surgery is mostly localized at the sternotomy site. To improve postoperative pain management a number of technics involving loco-regional anesthesia have been developed. The epidural analgesia is the gold standard but the risk of epidural hematoma with heparinization in this surgery avoids its utilization in clinical practice. The paravertebral block can be used equally but there is a risk of pneumothorax. The erector spinae plane block could be a solution as it is a more superficial block. It's efficacity was proven in thoracic and abdominal surgery, but literature is lacking in cardiac surgery. A bilateral erector spinae plane block after cardiac surgery could significantly reduce pain at rest and during mobilization, reduce opioids consumption, decrease postoperative complications, improve respiratory outcomes and improve patient comfort and satisfaction.

The main objective of this to study is to examine the efficacity of a single-shot bilateral erector spinae plane block on pain reduction during mobilization during the first 48 hours after cardiac surgery compared to a control group.

The primary outcome:

Pain scale at patient mobilization during the first postoperative 48 hours measured by numerical pain scale.

Study design:

Prospective, randomized, doubled-blinded, single-center controlled trial with two groups:

1. The ropivacaine group (42 patients): a bilateral erector spinae block will be performed after patient arrival in the intensive care unit before wake up from anesthesia with 20ml of Ropivacaine 2mg/ml bilaterally.
2. The control group (42 patients): a sham block will be performed bilaterally in the same conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo scheduled cardiac surgery with sternotomy for aortic or mitral valve replacement either by biological or mechanical prothesis, coronary arterial bypass surgery (CABG).
* Body Mass Index between 18,5 and 33kg/m² (extremity excluded)
* Patients who have given their consent according to the methods described in Title II of the book of the first Public Health Code
* Possession of Social Security insurance

Exclusion Criteria:

* Emergency surgery
* Approach by thoracotomy
* Heart transplant
* Aortic dissection or chirurgical act on ascending thoracic Aorta
* Redo surgery.
* Pregnant women
* Protected minors or adults
* Pre-existing psychiatric pathology including known states of opioid addiction
* Long-term opioid medication (>1month)
* Physical or intellectual inability to use a PCA
* Severe heart failure (ejection fraction less than 40% or PAH > 50 mmHg)
* Preoperative cardiogenic shock
* Severe preoperative chronic or acute renal failure with a creatinine clearance of less than 30 mL / min according to Cockroft's formula
* Known allergy or hypersensitivity to any of the study drugs or analgesia protocol (ropivacaine, paracetamol, opiates).
* Known allergy or hypersensitivity to any of excipients of the study drugs or analgesia protocol
* Refusal of the protocol

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change of pain score during cough | From patient awakening to 48 hours later (one evalution every 4 hours)
  Pain evaluation by a nurse with Numeric Rating Scale (with 0 = no pain; 10= maximum pain) during cough

SECONDARY OUTCOMES:
Change of pain score during patient tourn in the bed (lateralization) for nursing | From patient awakening to 48 hours later (one evalution every 4 hours)
  Pain score evaluation by a nurse with Numeric Rating Scale (with 0 = no pain; 10= maximum pain) during patient lateralization
Change of pain score during central venous pressure measuring | From patient awakening to 48 hours later (one evalution every 4 hours)
  Pain score evaluation by a nurse with Numeric Rating Scale (with 0 = no pain; 10= maximum pain) during patient lateralization
Change of sternal pain score at rest | From patient awakening to 48 hours later (one evalution every 4 hours)
  Pain score evaluation by a nurse with Numeric Rating Scale (with 0 = no pain; 10= maximum pain) during patient lateralization
Change of dorsal pain evaluation at rest | From patient awakening to 48 hours later (one evalution every 4 hours)
  Pain score evaluation by a nurse with Numeric Rating Scale (with 0 = no pain; 10= maximum pain) during patient lateralization
Opioid consumption | 48 hours after intervention
  Total opioid consumption since the awakening of the patient during 48 postoperative hours.
Satisfaction assessed by the Likert scale | 48 hours after intervention
  Subjective Assessment of pain management by the patient on a Likert scale going from 0 to 4 where 4 is excellent
Spirometry measure of forced vital capacity (FVC) | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the change of FVC by repeating spirometry during the hospital stay
Spirometry measure of forced expiratory volume in one second (FEV1) | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the change of FEV1 by repeating spirometry during the hospital stay
Spirometry measure of FEV1/FVC | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the change of FEV1/FVC by repeating spirometry during the hospital stay
Spirometry measure of peak expiratory flow (PEF) | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the change of PEF by repeating spirometry during the hospital stay
Spirometry measure of force expiratory flow 25% (FEF 25%), FEF 50%, FEF 75%, FEF 25-75% | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the change of FEF 25%, FEF 50%, FEF 75%, FEF 25-75% by repeating spirometry during the hospital stay
Diaphragmatic excursion | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the diaphragmatic excursion by repeating diaphragm echography during the hospital stay
Diaphragm thickness | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Assessment of the diaphragmatic thickness by repeating diaphragm echography during the hospital stay
Diaphragm thickening fraction | Up to 6 months after surgery (end of Hospital stay)
  Assessment of the diaphragmatic thickening fraction (%) by repeating diaphragm echography during the hospital stay
Digestive function | The day before surgery, the first or second day after surgery and the seventh day after surgery
  Time of recovery of normal bowel function. Beginning of oral feeding
Digestive function | Up to 6 months after surgery (end of Hospital stay)
  Time of recovery of normal bowel function.. Incidence of postoperative nausea and vomiting
Time of drain removal | Up to 6 months after surgery (end of Hospital stay)
  Time when the drain are removed of the patient
  Time when the drain are removed of the patient
Postoperative complications | Up to 1 month after surgery
  occurrence of postoperative respiratory, cardiac, renal, neurological, and infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Eljezi, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France